CLINICAL TRIAL: NCT01195038
Title: A Multicenter, Open-Label Study to Assess the Immunogenicity and Safety of a Booster Vaccination With a Recombinant H5N1 Influenza HA Vaccine in Healthy Young Adults Primed With a Two-Vaccination of a Recombinant H5N1 Influenza HA Vaccine
Brief Title: Immunogenicity and Safety Study of a Booster Vaccination With a Recombinant H5N1 Influenza HA Vaccine in Primed Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMN Pharma Inc. (Industry)
Responsible Party: UMN Pharma, Clinical Research Division
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JPIP501-01b
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Influenza
Keywords: Avian influenza, H5N1, pandemic, recombinant HA vaccine
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — FluBlok

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Recombinant Influenza HA Vaccine (H5N1) — one booster dose of 45 μg rHA derived from A/Indonesia/05/2005 strain
  Other Names: UMN-0501

SUMMARY:
The study is designed to assess the immunogenicity and safety of one booster vaccination with 45 μg of a recombinant H5N1 influenza (A/Indonesia/05/2005) HA vaccine in healthy young adults, previously primed with a two-vaccination of 3 different doses of a recombinant H5N1 influenza (A/Vietnam/1203/2004) HA vaccine in a priming study (JPIP501-01a, NCT00980447).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed a priming study (JPIP501-01a, NCT00980447)
* Male and female healthy adults
* Written informed consent obtained from the subject before study entry

Exclusion Criteria:

* History of H5N1 influenza or vaccination of other H5N1 influenza vaccines
* Clinically diagnosed cardiovascular, hematological, psychological, neurological, hepatic, renal, pulmonary (including asthma), endocrinological or gastrointestinal disorder
* Confirmed immune deficiency conditions, or diagnosed autoimmune diseases such as rheumatoid arthritis and systemic lupus erythematosus
* Severe allergic reactions or anaphylaxis to foods or drugs (including vaccines)
* Treatment with disallowed drugs including other study drugs
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 21 Years to 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving seroconversion 21 days after a booster vaccination, as measured by hemagglutination inhibition (HI) assay against H5N1 influenza viruses (A/Indonesia/05/2005 & A/Vietnam/1203/2004) | Day 21

SECONDARY OUTCOMES:
Percentage of subjects achieving seroprotection or significant increase in antibody titer on each blood sampling days after a booster vaccination, as measured by HI and microneutralization assays against the H5N1 influenza viruses | Days 7, 21
Incidence of adverse events including solicited local or systemic reactions until 21 days after a booster vaccination | 21 days

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - UMN Investigational Site, Osaka
  - UMN Investigational Site, Tokyo